CLINICAL TRIAL: NCT00232869
Title: A Clinical Investigation of the SIROlimus Coated Cordis SMART™ Nitinol Selfexpandable Stent for the Treatment of Obstructive Superficial Femoral Artery Disease.
Brief Title: A Study of the SMART Stent in the Treatment SFA Disease.
Acronym: SIROCCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EE00-02
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sirolimus Coated Cordis SMART™ nitinol selfexpandable stent
  Interventions: Device: drug-eluting stent
- 2 (Active Comparator): SMART™ bare-metal stent
  Interventions: Device: bare-metal stent

INTERVENTIONS:
Device: drug-eluting stent — Sirolimus Coated Cordis SMART™ nitinol selfexpandable stent
  Arms: 1
Device: bare-metal stent — SMART™ bare-metal stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and performance of the sirolimus coated Cordis SMART™ nitinol self expandable stent device and its delivery system in the treatment of obstructive superficial femoral artery (SFA) disease in reducing percent in-stent mean lumen diameter stenosis in de novo or restenotic native lesions as compared to the uncoated SMART™ stent.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, double blind, two-arm feasibility study evaluating the safety and performance of the sirolimus coated Cordis SMART™ nitinol self-expanding stent and delivery system as compared to the uncoated SMART™ stent and delivery system. It is anticipated that a total of 90 patients will be entered into the study. Patients will be randomized on a 1:1 basis of coated to uncoated stents.

Ninety (90) patients with de novo or restenotic native SFA lesions will be randomized to the Sirolimus Coated SMART™ nitinol self-expanding stent or to the uncoated (bare) SMART™ stent.

Patients will be followed for 24 months post-procedure, with all patients having duplex ultrasound and clinical assessments at discharge, 1, 6, 9, 18 and 24 months, angiography at 6 six months and plain X-ray at 18 months. This study will be conducted at nine investigational sites. (Protocol was amended where 56 additional patients were recruited and followed for up to 5 years.)

ELIGIBILITY:
Inclusion Criteria:

1. One superficial femoral artery presenting > 70% stenosis(es) or total occlusion
2. Symptomatic leg ischemia by Rutherford Classification (category 1, 2, 3 or 4)

Exclusion Criteria:

1. Tissue loss due to ischemic disease (Rutherford category 5 or 6).
2. Tandem lesion requiring non overlapping stents;

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2001-02; Primary Completion 2003-06 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
In-stent mean lumen diameter percent stenosis via quantitative angiography. | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan H Duda, MD, Principal Investigator — Tübingen - Germany
Locations (1):
- University Hospital, Tübingen, Germany

REFERENCES:
- [Result] Duda SH, Bosiers M, Lammer J, Scheinert D, Zeller T, Oliva V, Tielbeek A, Anderson J, Wiesinger B, Tepe G, Lansky A, Jaff MR, Mudde C, Tielemans H, Beregi JP. Drug-eluting and bare nitinol stents for the treatment of atherosclerotic lesions in the superficial femoral artery: long-term results from the SIROCCO trial. J Endovasc Ther. 2006 Dec;13(6):701-10. doi: 10.1583/05-1704.1. PMID 17154704